CLINICAL TRIAL: NCT05189652
Title: Investigation of the Effect of Myofascial Release Applied to Thoracolumbar Fascia on Flexibility, Muscular Endurance and Balance in Healthy Young Adults: A Pilot Study
Brief Title: Effect of Remote Myofascial Release on Lower Limb
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Collaborators: Akdeniz University (Other)
Responsible Party: Principal Investigator, UMMUHAN BAS ASLAN, Prof. Dr., Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Master Thesis
Record Dates: First submitted 2021-12-06; First posted 2022-01-12 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Flexibility; Balance; Muscular Endurance
MeSH Terms: interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Myofascial Release and Exercise Group (Experimental): Foam roller massage will be applied to the thoracolumbar posterior chain for participants in the myofascial release and exercise group. At the same time, balance training, squat exercises, reach forward with sitting and hamstring stretching exercises will be applied to this group for a period of four weeks. Before starting the exercise training programs, a 5 minute warm-up will be done. The first evaluation of the participants will be made before starting the 4-week program. Final assessments will be made within 2-3 days after the 4-week training ends. Evaluations will include flexibility measurements, muscular endurance measurements, balance evaluations.
  Interventions: Other: Myofascial Release and Exercise Group
- Exercise Group (Experimental): For the participants in the exercise group, the exercise program (balance training, squat exercises, reach forward with sitting and hamstring stretching exercises) will be applied 3 days a week for 4 weeks without any intervention to the thoracolumbar fascia. Before starting the exercise training programs, a 5 minute warm-up will be done. The first evaluation of the participants will be made before starting the 4-week program. Final assessments will be made within 2-3 days after the 4-week training ends. Evaluations will include flexibility measurements, muscular endurance measurements, balance evaluations.
  Interventions: Other: Exercise Group
- Control Group (No Intervention): Any myofascial release or exercise program will not be applied to the participants in the control group. The first evaluation of the participants will be made before other groups starting the 4-week program. Final assessments will be made within 2-3 days after the other groups 4-week training ends. Evaluations will include flexibility measurements, muscular endurance measurements, balance evaluations.

INTERVENTIONS:
Other: Myofascial Release and Exercise Group — The exercise program will be applied 3 days a week for 4 weeks. Participants will warm up by walking for 5 minutes before exercise. Stretching exercises - Reach forward with sitting and hamstring (3 reps*30 sec).
  First 2 weeks:
  Squat exercise (3 sets of 10 reps). Standing on one leg with knee flexed and hip-knee flexed at 90 degrees (30 seconds).
  Star Excursion balance training (2 rounds to be applied). Foam Roller massage will apply to thoracolumbar posterior chain (1 set of 30 seconds will be applied with a rolling period of 2-4 seconds).
  Last 2 weeks:
  Squat exercise (3 sets of 15 reps). Standing on one leg with knee flexed and hip-knee flexed at 90 degrees (40 seconds).
  Star Excursion balance training (3 rounds to be applied). Foam Roller massage will apply to thoracolumbar posterior chain (2 sets of 30 seconds will be applied to each area with a rolling period of 2-4 seconds).
  Arms: Myofascial Release and Exercise Group
Other: Exercise Group — The exercise program will be applied 3 days a week for 4 weeks. Participants will warm up by walking for 5 minutes before exercise. Stretching exercises- Reach forward with sitting and hamstring (3 reps*30 sec).
  First 2 weeks:
  Squat exercise (3 sets of 10 reps). Standing on one leg with knee flexed and hip-knee flexed at 90 degrees (30 seconds).
  Star Excursion balance training (2 rounds to be applied).
  Last 2 weeks:
  Squat exercise (3 sets of 15 reps). Standing on one leg with knee flexed and hip-knee flexed at 90 degrees (40 seconds).
  Star Excursion balance training (3 rounds to be applied).
  Arms: Exercise Group

SUMMARY:
In general, the strength training on unstable surfaces has a positive impact on strength performance, power and stability compared to not training. As described above, previous studies have shown that self-myofascial release has a positive effect by improving flexibility, but its effect on balance is still debated.

Myofascia contains numerous sensory nerves related to proprioceptive and mechanical receptors such as Golgi receptors or Pacini receptors. Therefore, the pressure applied during the self-myofascial release intervention can stimulate these mechanoreceptors and enhance the proprioceptive information integrated by the central nervous system to adjust the activation level of motor units. The aim of this study is to examine the effects of myofascial release applied to the thoracolumbar fascia on flexibility, muscular endurance and balance in healthy young adults.

DETAILED DESCRIPTION:
Fascia, muscles, bones, organs, nerves, it refers to all fibrous ligament tissue under stress that both encompasses and surrounds blood vessels and other structures, and stretches from head to foot in a continuous, three-dimensional network. Fascia is the most sensitive and vital structure in our bodies, linked to systems in the whole body, as vital as blood. This structure is a system of a single tissue fiber that is located directly below the skin. Fascia stretches through the whole body in lines for a locked-in feel. Thoracolumbar fascia (TLF) is an important structure that connects the lower extremity to the gluteus maximum and the upper extremity to the latissimus dorsi. The thoracolumbar fascia allows trunk stabilization in kinetic chain activities including movements such as throwing. The thoracolumbar fascia surrounds different trunk muscles, such as the multifidus, erector spines, and quadratus lumborum and provides support when these muscles contract. It also attaches to the internal oblique, transversus abdominis, latissimus dorsi aponeurosis and serratus anterior inferior muscle. Contraction of these muscles increases tension along the fascia and stabilizes the trunk by providing 3-dimensional support to the lumbar spine.

The fasciae of the transversus abdominis, internal oblique and quadratus lumborum muscles are surrounded by the thoracolumbar fascia. The transversus abdominis muscle stabilizes the lumbo-pelvic region by stretching the thoracolumbar fascia and increasing intra-abdominal pressure. Thoracolumbar fascia, lower extremity and upper extremity acts as part of a pulley around the body, which provides a connection. Fascia disorders are often associated with adaptive misuse of muscles. For this reason, myofascial treatment is usually supported by appropriate exercises that the person will do. In this way, while creating a conscious awareness of the normal function of the patient in that muscle, it can reprogram the brainstem to incorporate the newly restored full-scale muscle capacity into the patient's daily activities.

In recent years, the popularity of training has increased with the foam roller, which is one of the myofascial treatment methods. Foam roller massage is a relatively new technique and a common form of self-myofascial training performed by participants themselves and not by a clinician. The foam roller is a solid foam cylinder available in different stiffness and size. Athletes or patients are encouraged to rotate their body weights to operate each muscle group and loosen tight areas of the muscle. A possible effect is better moisturizing of tissues. While applying the foam roller massage, the soft tissue is squeezed like a sponge and then wetted with liquid, which improves the movement between the different layers of the fascia. This method, which affects the muscle and myofascial structures by increasing the compatibility and extensibility of the fascia, reduces passive muscle stiffness. It can also reduce delayed onset muscle soreness after intense exercise. Self-myofascial release has been shown to provide a wide range of positive gains in physical performance. The best-known positive effect of self-myofascial release is a gain in flexibility as assessed by increased range of motion in sports and rehabilitation contexts. Scientifically, many positive effects of foam roller massage are assumed, but in most cases unproven. Most studies of self-myofascial release techniques address the acute effects, while there is limited clinical research on the training effects of foam roller massage. The sample will be adults between the ages of 18-40. Investigators will announce the research via social media and invite volunteers to work. Participants who are willing to participate will be explained the study and participants who agree to participate and who meet the work criteria will be included in the study. Participants will be divided into 3 groups as Myofascial Release and Exercise Group, Exercise Group, and Control Group using the computerized randomization method. Since the study is pilot operation, no power analysis has been performed to determine the sample size. Investigators aim to have at least 12 people in each study group. The first evaluation of the participants will be made before starting the 4-week program. Final assessments will be made within 2-3 days after the 4-week training ends. Evaluations will include flexibility measurements, muscular endurance measurements, balance evaluations. The study will have a single-blind design. The investigator making the evaluation will not know which group the participant is in.

ELIGIBILITY:
Inclusion Criteria:

* be between the ages of 18-40
* Volunteer

Exclusion Criteria:

* To have exercised regularly for the last 6 months
* Injury to the lower extremity in the last 6 months
* Having the condition in which the application of myofascial release is contraindicated
* Orthopedic, neurological, endocrine, vascular, etc. to prevent exercise structure having diseases

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-05-24 (Actual)

PRIMARY OUTCOMES:
Personal informations | 4 weeks
  Personal information questionnaire: The gender of the participants will be recorded by the investigator by ticking one of the male/female options. In the data analysis, the gender distribution of the participants will be expressed as a percentage.
Personal informations | 4 weeks
  Personal information questionnaire: 'How many years has your education life been?' the survey question will be asked and the length of time in the answer received by asking the question will be recorded by the investigator as the year. In the data analysis, the years of education of the participants will be expressed as the average of years.
Personal informations | 4 weeks
  Personal information questionnaire: Profession of the participants, 'Which profession do you do?' the answer received by asking the survey question will be recorded by the investigator. In the data analysis, the professions of the participants will be expressed as a percentage.
Personal informations | 4 weeks
  Personal information questionnaire: 'How long have you been doing your profession?' survey question will be asked. The length of time the participants work in the profession will be recorded by the investigator as the year. In the data analysis, the years of working time in profession of the participants will be expressed as the average of years.
Clinical status | 4 weeks
  Clinical status questionnaire: The age of the participants is, 'How old are you?' the answers received by asking the survey question will be recorded by the investigator as the year. In the data analysis, the ages of the participants will be expressed as the average of the years.
Clinical status | 4 weeks
  Height: Participants' height in cm will be recorded by the investigator.
Clinical status | 4 weeks
  Weight: Participants' weight in kg will be recorded by the investigator.
Clinical status | 4 weeks
  BMI: Participants' body mass index in kg/m^2 will be recorded by the investigator.
Clinical status | 4 weeks
  Clinical status questionnaire: To identify the participants' dominant lower extremity, when the participants are given the 'Jump on one foot' command, the preferred foot will be marked as the right or left extremity by the investigator. In the data analysis, the dominant extremities of the participants will be expressed as a percentage.
Clinical status | 4 weeks
  Clinical status questionnaire: The survey question 'Did you exercised regularly at least 2 days a week during the last 6 months' will be asked to the participants. Yes or no answers will be recorded by the investigator.
Clinical status | 4 weeks
  Clinical status questionnaire: In order to determine the smoking habits of the participants, the survey question 'Do you smoke?' will be asked and one of the smoker/non-smoker options will be marked by the investigator. In the data analysis, the smoking of the participants will be expressed as a percentage.
Flexibility measurements | 4 weeks
  Sit and Reach Test: A standard sit and reach box will be placed on the floor. Participants will be asked to sit on the floor on a flat surface and rest their bare feet flat on the test bench. Afterwards, participants will be asked to hold for a second or two at the last point, extending their torso forward as far as participants can reach, with the arms and fingers stretched and straight. For data analysis, each measurement will be repeated 2 times by the investigator. A ruler will be used as a measuring tool and the measurement result will be recorded in cm.
Flexibility measurements | 4 weeks
  Active Knee Extension Test: Participants will lie in the supine position with the hip joint and knee joint in 90 degrees flexion and the other knee will be kept flat on the ground. The participant will be asked to straighten the knee of the evaluated side as much as possible without disturbing the hip joint angle. At the last possible point, the degree of knee flexion will be measured by the investigator with a goniometer. Each measurement will be repeated 2 times for data analysis.
Muscular endurance measurements | 4 weeks
  1 Minute Sit to Stand Test: Participants will get up and sit in a chair without an armrest as many times as possible in 1 minute. The chair will be adjusted so that the angle of the knee joints is approximately 90° while sitting. During the test, participants will be asked to keep feet parallel and hands on waists to avoid using arms to assist with movement. Participants will be instructed to stand up when bringing knees to full extension and to touch the chair with hips while sitting. Participants will be instructed to do as many sit to stand repetitions as possible in 1 minute by the investigator. Participants will be informed with 15 seconds remaining but will not be motivated during the test. The number of complete and correct sit-to-stand cycles after 1 minute will be recorded by the investigator for analysis.
Static Balance | 4 weeks
  One-leg Standing Test: The duration of standing by reducing the support surface of the participants and maintaining balance on one leg with eyes open and closed will be recorded by the investigator. A stopwatch will be used as a measurement tool. The time from the moment the participants starts to stand on one leg until he loses his balance will be recorded in seconds. The test will be terminated if the participants can stand on one leg for 60 seconds without losing balance.
Dynamic Balance | 4 weeks
  Star Excursion Balance Test: A star shape will be drawn on the ground with a total of 8 directions at an angle of 45 degrees. Participants will be asked to reach these directions according to the predetermined protocol and the distance reached by the participants will be recorded by the investigator in cm. Before the application, the participants will be given a rest period of 180 seconds to familiarize themselves with the test and 120 seconds between applications. In addition, 5 seconds will be given by the researchers between each stretch so that participants can stand on good feet. In order to normalize the data, the leg length of the participants will be measured in cm between spina iliaca anterior superior-medial malleolus and recorded by the investigator. A tape measure will be used as a measuring tool. The measurement results will be recorded by the investigator in cm. Each measurement will be repeated 3 times for data analysis.
Fatigue | 4 weeks
  Modified Borg Fatigue Scale: The Modified Borg Scale will be used to assess the level of effort reported by participants during physical exercise. Participants will report perceived fatigue immediately after each exercise session on this scale from zero to ten (0-10). In this way, the intensity of the exercise will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Atacan Tonak, Asst. Prof. Dr., Principal Investigator — Akdeniz University; Hatice Ozdemir, PT, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Individual Participant Data Set — https://doi.org/10.2478/hukin-2020-0043 — Zhang, Q., Trama, R., Fouré, A., & Hautier, C. A. (2020). The Immediate Effects of Self-Myofacial Release on Flexibility, Jump Performance and Dynamic Balance Ability. Journal of human kinetics, 75, 139-148.